CLINICAL TRIAL: NCT07088952
Title: Triggering Ovulation at Follicle Size Smaller or Larger Than 17mm in a Modified Natural Cycle
Acronym: 17FET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2310-SEV-02-MF
Record Dates: First submitted 2025-06-17; First posted 2025-07-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Embryo Transfer
Keywords: Natural Cycle; Frozen Embryo Transfer; Follicle Size; Pregnancy; Implantation

STUDY DESIGN:
Intervention Model Description: Prospective open randomized parallel group 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Trigger indicated as per standard clinical practice at folicular diameter of at least 17mm
- Early trigger (Experimental): Trigger indicated at folicular diameter smaller than standard clinical practice
  Interventions: Procedure: Trigger at smaller folicular size

INTERVENTIONS:
Procedure: Trigger at smaller folicular size — Trigger indicated at folicular diameter smaller than standard clinical practice, from 13mm to 16.9mm
  Arms: Early trigger

SUMMARY:
The rise in frozen embryo transfer (FET) cycles within assisted reproductive technology (ART) has sparked the need to refine endometrial preparation protocols. The switch from hormone replacement cycles (HRT) to natural cycles, poses scheduling challenges onto laboratories, doctors and patients. The modified natural cycle (mNC), offering more precision for scheduling, shows promise but lacks comprehensive data on the potential flexibility of triggering criteria that may allow to control timing in a wider range.

This prospective randomized study seeks to address this knowledge gap by evaluating the non-inferiority of triggering ovulation in mNC with follicle diameters of 13-16.9mm compared to the conventional 17-22mm.

The study aims to enhance the understanding of the impact of follicle size at ovulation in reproductive outcomes, optimize FET treatments providing a more flexible mNC protocol, and improve patient care in ART clinics.

ELIGIBILITY:
Inclusion Criteria:

* At least one expanded blastocyst (regardless of its quality)
* Spontaneous menstrual cycles
* Consent to undergo frozen embryo transfer in a modified natural cycle

Exclusion Criteria:

* Abnormal uterine cavity
* Fluid in endometrial cavity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 572 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | From embryo transfer up to 2 weeks later
  Rate of positive pregnancies over total transfers performed, according to beta-test result

SECONDARY OUTCOMES:
Implantation rate | up to 8 weeks of gestational age
  Implantation rate, defined as number of gestational sacs per embryos transferred
Cancelation rate | Perioperative/Periprocedural
  Number of cancelled embryo transfers per initiated endometrial preparation cycles. Transfer canceling implies end of study.
Miscarriage rate | From embryo transfer to delivery, up to 40 weeks
  Number of miscarriages of any type registered after transfer during the study, per total number of transfers performed

CONTACTS AND LOCATIONS:
Locations (1):
- Vida Recoletas Sevilla, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.